CLINICAL TRIAL: NCT01549899
Title: Comparing Internet and In-Person Brief Cognitive Behavioral Therapy of Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel J. Taylor, Ph.D. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); C.R.Darnall Army Medical Center (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor-Investigator, Daniel J. Taylor, Ph.D., Professor, University of North Texas, Denton, TX
Organization: University of North Texas, Denton, TX (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-10-1-0828; PT090525 (Other: CDMRP)
Record Dates: First submitted 2012-02-04; First posted 2012-03-09 (Estimated); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive; Behavioral; Therapy; Internet; Depression; Substance Use; Post-Tramatic Stress Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Behavior; Depression; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- In-person CBT of Insomnia (Active Comparator): CBTi consisted of 6 weekly 60-minute sessions and included identical informational material. The treatments contained the following efficacious and commonly used modules of cognitive behavioral treatments for insomnia: Stimulus Control, Sleep Restriction, Sleep Hygiene, Relaxation Training, Cognitive Restructuring.
  Interventions: Behavioral: In-person Cognitive Behavioral Therapy of Insomnia
- Internet CBT of Insomnia (Active Comparator): The I-CBTi protocol was developed by the National Center for Telehealth and Technology with the first author (DJT) serving as the subject matter expert, and administered on the afterdeployment.org website. The information and instructions for I-CBTi were identical to in-person CBTi; however, their mode of delivery in I-CBTi is considerably different due to the constraints of its automated, online format. The lessons were presented as audio recordings accompanied by visual graphics and animations and several lessons, had interactive components such as games, quizzes, and prompts for participants to schedule healthy sleep habits.
  Interventions: Behavioral: Internet Cognitive Behavioral Therapy of Insomnia
- Minimal Contact (No Intervention): Those assigned to the MC control group will be asked to not work with another therapist or seek additional treatment for insomnia-related difficulties during the 6-week MC period. They will be called every other week to monitor their status and to provide support as needed. The calls will be limited to 10-15 minutes. MC participants will also be given contact information to use in case of worsening of symptoms or increasing distress. At the end of six weeks, they will complete the baseline assessments again, which will serve as the post-treatment assessment for the MC period. They will then be randomly assigned to either the CBTi or ICBTi groups.

INTERVENTIONS:
Behavioral: In-person Cognitive Behavioral Therapy of Insomnia — In-person CBTi was be provided by a master's or doctoral level mental health counselor (e.g., social worker or psychologist). This treatment consisted of 6-sessions and included the same efficacious and commonly used modules of CBTi (i.e., sleep education & hygiene, stimulus control, progressive muscle relaxation, sleep restriction, and cognitive therapy).
  Arms: In-person CBT of Insomnia
Behavioral: Internet Cognitive Behavioral Therapy of Insomnia — The ICBTi treatment is an online protocol developed by the National Center for Telehealth and Technology, with the PI (DJT) as the subject matter expert. The treatment consists of the same components as the in-person CBTi, but their mode of delivery was considerably different due to the constraints of its automated, online format. Each of the six ICBTi sessions was divided into lessons covering different aspects of each of the components. The lessons were presented as audio recordings accompanied by visual graphics and animations. For several lessons, interactive components were included, such as games, quizzes, and prompts for participants to schedule healthy sleep habits.
  Arms: Internet CBT of Insomnia

SUMMARY:
The objective of this study is to directly compare 6 sessions of in-person and Internet administered Cognitive-Behavior Therapy for Insomnia (CBTi) to a Minimal Contact control (MC), within an active duty military population to determine the comparative benefits of these interventions on improvement in sleep as well as domains strongly related to insomnia such as depression, substance abuse, and PTSD symptoms. A total of 189 military personnel with chronic insomnia, aged 18-65, will be recruited and randomized to receive 6-sessions (over 6 weeks) of CBTi (n=77), ICBTi (n=35), or a MC control (n=77) condition. The investigators will compare these three groups on subjective and objective measures of sleep. The CBTi and MC control groups will be compared on other variables of interest (e.g., depression, substance abuse, and PTSD symptoms) and predictors of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Insomnia as defined by Research Diagnostic Criteria (RDC) criteria41 Complaint of > 3 months (chronic insomnia) of disturbed sleep >3 nights/week (severe insomnia) as defined by at least one of the following as assessed by sleep diaries: Sleep Onset Latency of >30 min (initial insomnia) and/or Wake After Sleep-Onset of >30 min (middle insomnia) and/or Early Morning Awakening of >30 min before the desired wakeup time (late insomnia) and Sleep Efficiency < 85%
* Active Duty military member stationed at Fort Hood as assessed by self-report.
* History of having deployed in support of OIF or OEF as assessed by self-report. • Stable on psychotropic and/or hypnotic medications for at least one month as assessed by self-report and review of medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Taylor, Ph.D., Principal Investigator — University of North Texas Health Science Center
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States

REFERENCES:
- [Background] Taylor DJ, Wilkerson AK, Pruiksma KE, Williams JM, Ruggero CJ, Hale W, Mintz J, Organek KM, Nicholson KL, Litz BT, Young-McCaughan S, Dondanville KA, Borah EV, Brundige A, Peterson AL; STRONG STAR Consortium. Reliability of the Structured Clinical Interview for DSM-5 Sleep Disorders Module. J Clin Sleep Med. 2018 Mar 15;14(3):459-464. doi: 10.5664/jcsm.7000. PMID 29458705
- [Background] Peterson AL, Young-McCaughan S, Roache JD, Mintz J, Litz BT, Williamson DE, Resick PA, Foa EB, McGeary DD, Dondanville KA, Taylor DJ, Wachen JS, Fox PT, Bryan CJ, McLean CP, Pruiksma KE, Yarvis JS, Niles BL, Abdallah CG, Averill LA, Back SE, Baker MT, Blount TH, Borah AM, Borah EV, Brock MS, Brown LA, Burg MM, Cigrang JA, DeBeer BB, DeVoe ER, Fina BA, Flanagan JC, Fredman SJ, Gardner CL, Gatchel RR, Goodie JL, Gueorguieva R, Higgs JB, Jacoby VM, Kelly KM, Krystal JH, Lapiz-Bluhm MD, Lopez-Roca AL, Marx BP, Maurer DM, McDevitt-Murphy ME, McGeary CA, Meyer EC, Miles SR, Monson CM, Morilak DA, Moring JC, Mysliwiec V, Nicholson KL, Rauch SAM, Riggs DS, Rosen CS, Rudd MD, Schobitz RP, Schrader CC, Shinn AM, Shiroma PR, Sloan DM, Stern SL, Strong R, Vannoy SD, Young KA, Keane TM; STRONG STAR Consortium and the Consortium to Alleviate PTSD. STRONG STAR and the Consortium to Alleviate PTSD: Shaping the future of combat PTSD and related conditions in military and veteran populations. Contemp Clin Trials. 2021 Nov;110:106583. doi: 10.1016/j.cct.2021.106583. Epub 2021 Sep 29. PMID 34600107
- [Background] Brown LA, Zang Y, Benhamou K, Taylor DJ, Bryan CJ, Yarvis JS, Dondanville KA, Litz BT, Mintz J, Roache JD, Pruiksma KE, Fina BA, Young-McCaughan S, Peterson AL, Foa EB; STRONG STAR Consortium. Mediation of suicide ideation in prolonged exposure therapy for posttraumatic stress disorder. Behav Res Ther. 2019 Aug;119:103409. doi: 10.1016/j.brat.2019.103409. Epub 2019 May 23. PMID 31176888
- [Background] Brown LA, Bryan CJ, Butner JE, Tabares JV, Young-McCaughan S, Hale WJ, Fina BA, Foa EB, Resick PA, Taylor DJ, Coon H, Williamson DE, Dondanville KA, Borah EV, McLean CP, Wachen JS, Pruiksma KE, Hernandez AM, Litz BT, Mintz J, Yarvis JS, Borah AM, Nicholson KL, Maurer DM, Kelly KM, Peterson AL; STRONG STAR Consortium. Identifying suicidal subtypes and dynamic indicators of increasing and decreasing suicide risk in active duty military personnel: Study protocol. Contemp Clin Trials Commun. 2021 Feb 16;21:100752. doi: 10.1016/j.conctc.2021.100752. eCollection 2021 Mar. PMID 33748530
- [Background] Ben Barnes J, Presseau C, Jordan AH, Kline NK, Young-McCaughan S, Keane TM, Peterson AL, Litz BT; the Consortium to Alleviate PTSD. Common Data Elements in the Assessment of Military-Related PTSD Research Applied in the Consortium to Alleviate PTSD. Mil Med. 2019 May 1;184(5-6):e218-e226. doi: 10.1093/milmed/usy226. PMID 30252077
- [Result] Taylor DJ, Peterson AL, Pruiksma KE, Hale WJ, Young-McCaughan S, Wilkerson A, Nicholson K, Litz BT, Dondanville KA, Roache JD, Borah EV, Brundige A, Mintz J; STRONG STAR Consortium. Impact of cognitive behavioral therapy for insomnia disorder on sleep and comorbid symptoms in military personnel: a randomized clinical trial. Sleep. 2018 Jun 1;41(6). doi: 10.1093/sleep/zsy069. PMID 29618098
- [Result] Taylor DJ, Peterson AL, Pruiksma KE, Young-McCaughan S, Nicholson K, Mintz J; STRONG STAR Consortium. Internet and In-Person Cognitive Behavioral Therapy for Insomnia in Military Personnel: A Randomized Clinical Trial. Sleep. 2017 Jun 1;40(6). doi: 10.1093/sleep/zsx075. PMID 28472528
- [Result] Pruiksma KE, Hale WJ, Mintz J, Peterson AL, Young-McCaughan S, Wilkerson A, Nicholson K, Dondanville KA, Fina BA, Borah EV, Roache JD, Litz BT, Bryan CJ, Taylor DJ; STRONG STAR Consortium. Predictors of Cognitive Behavioral Therapy for Insomnia (CBTi) Outcomes in Active-Duty U.S. Army Personnel. Behav Ther. 2020 Jul;51(4):522-534. doi: 10.1016/j.beth.2020.02.001. Epub 2020 Feb 14. PMID 32586427

RESULTS

PARTICIPANT FLOW:
Groups:
- Internet CBT of Insomnia: Internet Cognitive Behavioral Therapy of Insomnia: The ICBTi treatment is an online protocol developed by the National Center for Telehealth and Technology, with the PI (DJT) as the subject matter expert. The treatment consists of the same components as the in-person CBTi, but their mode of delivery was considerably different due to the constraints of its automated, online format. Each of the 6 ICBTi sessions was divided into lessons covering different aspects of each of the components. The lessons were presented as audio recordings accompanied by visual graphics and animations. For several lessons, interactive components were included, such as games, quizzes, and prompts for participants to schedule healthy sleep habits.
Period: Overall Study
Arm/Group | In-person CBT of Insomnia | Internet CBT of Insomnia | Minimal Contact
Started | 75 | 34 (Are discontinued at n = 34 due to irreparable technical issues with internet CBTi.) | 76
Completed | 63 | 27 | 68
Not Completed | 12 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-person CBT of Insomnia | Internet CBT of Insomnia | Minimal Contact | Total
Number analyzed (Participants) | 75 | 34 | 76 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.21 (7.18) | 34.53 (8.27) | 32.67 (7.97) | 32.44 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 14 | 33
  Male | 62 | 28 | 62 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 19 | 8 | 27 | 54
  Hispanic | 14 | 3 | 12 | 29
  Caucasian | 39 | 21 | 30 | 90
  Other | 3 | 2 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Sleep Diary Sleep Efficiency
Description: Provides daily self-reports of bedtime, time to fall asleep, middle of the night awakenings, and time out of bed. These data will be aggregated to determine self-reported sleep efficiency (i.e., total sleep time/time in bed X 100). Other variable to be extracted will include total sleep time and total wake time.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Measure: Mean (Standard Error); unit: Percentage Total Sleep Time/Time in Bed
Groups:
- Internet CBT of Insomnia: The I-CBTi protocol was developed by the National Center for Telehealth and Technology with the first author (DJT) serving as the subject matter expert, and administered on the afterdeployment.org website. The information and instructions for I-CBTi were identical to in-person CBTi; however, their mode of delivery in I-CBTi is considerably different due to the constraints of its automated, online format. The lessons were presented as audio recordings accompanied by visual graphics and animations and several lessons, had interactive components such as games, quizzes, and prompts for participants to schedule healthy sleep habits.
  Internet Cognitive Behavioral Therapy of Insomnia: The ICBTi treatment is an online protocol developed by the National Center for Telehealth and Technology, with the PI (DJT) as the subject matter expert. The treatment consists of the same components as the in-person CBTi, but their mode of delivery was considerably different due to the constraints of its aut
Arm/Group | In-person CBT of Insomnia | Internet CBT of Insomnia | Minimal Contact
Number analyzed (Participants) | 33 | 34 | 33
Percentage Total Sleep Time/Time in Bed
  Baseline | 73.2 (2.2) | 72.5 (2.1) | 72.9 (2.2)
  Post-treatment | 84.5 (2.2) | 79.4 (2.4) | 73.1 (2.3)

2. Secondary Outcome: Beck Depression Inventory II
Description: Measure of self-reported depression symptoms.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Substance Use
Description: Self-reported use of sleep medications, caffeine, and nicotine obtained during the interview and on sleep diaries.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Actigraphy
Description: A wrist worn accelerometer that measures activity level and then uses validated algorithms to determine objectively daily bedtime, time to fall asleep, middle of the night awakenings, and time out of bed. These data will be aggregated to determine objective sleep efficiency (i.e., total sleep time/time in bed X 100). Other variable to be extracted will include total sleep time and total wake time.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

5. Secondary Outcome: PTSD Check List-Military
Description: Measures self-reported Post-Traumatic Stress Disorders symptoms in military personnel.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Beck Anxiety Inventory
Description: Self-report measure of anxiety symptoms
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

7. Secondary Outcome: Insomnia Severity Index
Description: Self-report insomnia symptoms.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

8. Secondary Outcome: Epworth Sleepiness Scale
Description: Self-report daytime sleepiness.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

9. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep Scale
Description: Self-reported beliefs and attitudes about sleep.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

10. Secondary Outcome: Multidimensional Fatigue Inventory
Description: Self-reported fatigue symptoms across multiple dimensions.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

11. Secondary Outcome: Veterans Rand 12-Item Health Survey
Description: Self-reported quality of life and health.
Time Frame: Change from Baseline to Post-Treatment and 6 month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time frame was from Baseline to Post-treatment. However, the collection rate was different among groups.
Description: The In-Person were asked during their weekly visits by a therapist. The Internet and Minimal Contact had every other week phone calls, but participants often did not answer or respond because they were active duty military and at their jobs for the Army. Thus, the collection rate was ~>66% more often in the In-person than other two groups.
Arm/Group | In-person CBT of Insomnia | Internet CBT of Insomnia | Minimal Contact
All-Cause Mortality (participants affected / at risk) | 52/75 | 8/34 | 10/76
Serious Adverse Events (participants affected / at risk) | 5/75 | 0/34 | 1/76
Other Adverse Events (participants affected / at risk) | 47/75 | 8/34 | 9/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-person CBT of Insomnia (N=75) | Internet CBT of Insomnia (N=34) | Minimal Contact (N=76)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Accident (General disorders) | 3 (3) | 0 (0) | 1 (1) — Participant had an accident outside of the study. Went to ER, not hospitalized.
Alcohol-Detox (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Participant was admitted to 28-day inpatient program.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-person CBT of Insomnia (N=75) | Internet CBT of Insomnia (N=34) | Minimal Contact (N=76)
Headache, Migraine (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anxiety, Panic (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep Walking (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory, Blackout (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cold/ flu (Infections and infestations) | 11 (11) | 1 (1) | 3 (3)
Allergies (General disorders) | 5 (5) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain, Arthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) | 0 (0)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Rash (General disorders) | 3 (3) | 1 (1) | 1 (1)
GI disturbance (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Visual Disturbance (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Other (General disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No